CLINICAL TRIAL: NCT06414252
Title: Functional Physiological, Psychological and Biochemical Reactivity to Social Evaluated Cold Pressor Test in Hereditary Angioedema Patients
Brief Title: Social Evaluated Cold Pressor Test in Hereditary Angioedema Patients
Acronym: FROSEN
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 2774CE
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; Autonomic nervous system; Cold pressor test; Stress; Body appreciation; Rare disease
MeSH Terms: conditions — Angioedemas, Hereditary; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hereditary angioedema: Patients with documented diagnosis of hereditary angioedema due to C1 inhibitor deficiency and aged between 18 and 65 years.
- Healthy individuals: Healthy individuals with an age between 18 and 65 and matched with patients with hereditary angioedema by age and gender.

SUMMARY:
This study aims to evaluate the differences in objective and subjective stress responses between patients with hereditary angioedema and healthy individuals to a stress-induced challenge like socially-evaluated cold pressure test. The study also investigates the role of psychological variables in influencing the stress response.

DETAILED DESCRIPTION:
Stressful encounters, ranging from daily hassles to major life events, are ubiquitous in our everyday lives and are often responsible for significant changes in affective and cognitive processes. In various physical diseases, including hereditary angioedema (HAE) due to C1 inhibitor deficiency, stressful events are also frequently reported by patients to trigger acute attacks. These include physical stress (such as injury, pain, viral infections, medical and dental procedures, and surgery) and mental stress (including stress from life events and school or work, clinical depression, and anxiety), or stress originating from the disease itself, especially if the disease is characterized by an unpredictable nature like HEA that directly impacts patients' choices in everyday life. Available literature related to the link between HAE and stress is limited and mainly focused on the patients' narratives. Self-reported data suggested that the main HAE trigger seems to be stress, followed by physical trauma. These observations suggest analyzing the perceived psychological effects consequent to stress exposure together with biochemical and physiological responses. The effect of stress could be systematically examined in a laboratory environment using a standardized protocol that reliably induces stress and activates major stress responses in experimental contexts. A reliable test to induce stress in HAE patients combining these two aspects may be the Socially Evaluated Cold Pressor Test (SECPT). SECPT is an extension of the classical Cold Pressor Test, in which participants immerse one of their hands in ice water with socio-evaluative elements, and has been proven to be a highly efficient tool for experimental stress induction in humans. Adding social-evaluative elements to the original physical stress boosted the cortisol response, making the SECPT a well-established standard protocol in human stress research that may represent an efficient alternative to other established protocols, such as the Trier Social Stress Test, a 'gold standard' in the field. A recent review confirmed that exposure to the SECPT leads to changes in subjective feeling, and triggers a significant sharp increase in systolic and diastolic blood pressure. The present study aims to evaluate objective and subjective stress responses between HAE patients and healthy controls due to SECPT. Moreover, as secondary aims, the study wants to investigate if the presence of anxiety and depressive symptoms, as well as body appreciation, trust in the body, pain catastrophizing, pain interference, and pain intensity, affect or mediate stress response in patients and healthy subjects similarly or differently.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of hereditary angioedema due to C1 inhibitor deficiency aged between 18 and 65 years (for the group of patients)

Exclusion Criteria:

* Any type of chronic disease requiring chronic treatment (i.e. hypertension, previous myocardial infarction, diabetes, chronic heart failure, autoimmune disease, neurodegenerative disease)
* Active acute disease;
* Sars-Cov2 infection in the previous 3 months.
* An acute attack experienced within the previous week and within 72 hours after the registration (a posteriori exclusion).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The group of patients with hereditary angioedema were recruited during an out-patient visit in a tertiary care center. The group of healthy individuals were volunteers recruited from community.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Heart rate | Baseline
  Changes in the heart rate (beats per minute) from resting to SECPT condition
Systolic arterial pressure | Baseline
  Changes in the systolic blood pressure (mmHg) from resting to SECPT condition
Diastolic arterial pressure | Baseline
  Changes in the systolic blood pressure (mmHg) from resting to SECPT condition
Visual Analogue Scale of perceived stress | Baseline
  Changes in the perceived stress due to SECP. Scores ranges from 0 (no stress) to 100 (worst stress possible)
Concentration of inflammatory cytokines | Baseline
  Changes in the concentration of inflammatory cytokines (pg/ml) due to SECPT
Concentration of plasma cathecolamines | Baseline
  Changes in the concentration of plasma cathecolamines (pg/ml) due to SECPT

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline
  A 14-item questionnaire subdivided in two subscales to measure anxiety and depression. Scores for each subscale ranges from 0 (absence of symptoms) to 21 (significant symptoms)
Perceived Stress Scale (PSS-10) | Baseline
  A 10-item questionnaire to measure stress levels related to the perception of unpredicable, uncontrollable, and overloading nature of life. Scores ranges from 0 (low levels) to 40 (high levels).
Multidimensional Assessment of Interoceptive Awareness Version 1 | Baseline
  A 32-item questionnaire to measure Interoceptive Awareness. Scores ranges from 0 (low interoceptive awareness) to 160 (high interoceptive awareness).
Body Appreciation Scale-2 (BAS-2) | Baseline
  A 10-item questionnaire to measure appreciation. Scores ranges from 10 (low body appreciation) to 50 (high body appreciation).
Functionality Appreciation Scale (FAS) | Baseline
  A 7-item questionnaire to measure body appreciation. Scores ranges from 0 (low functionality appreciation) to 35 (high functionality appreciation)
Pain Catastrophizing Scale (PCS) | Baseline
  A 13-item questionnaire to measure pain-related catastrophizing. Scores ranges from 0 (low catastrophizing ) to 52 (high catastrophizing).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Milan, Italy

REFERENCES:
- [Derived] De Maria B, Ranucci L, Gino C, Cesoni Marcelli A, Zingale LC, Zulueta A, Dalla Vecchia LA, Gorini A, Perego F. Functional physiological, psychological, and biochemical reactivity to socially evaluated cold pressor test in hereditary angioedema patients (FRoSEn). Front Immunol. 2026 Jan 7;16:1736589. doi: 10.3389/fimmu.2025.1736589. eCollection 2025. PMID 41573571